CLINICAL TRIAL: NCT04362371
Title: Post Marketing Follow Up Study To Evaluate Performance, Safety And Quality Of Life In Late Menopausal Transition And Post-Menopausal Women Treated With The Medical Device Ainara® Vaginal Gel, For Vaginal Dryness For 6 Months
Brief Title: Post Marketing Follow Up Study To Evaluate Performance Safety Quality of Menopausal Transition Women Treated With Ainara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS/18/AINARA/03
Record Dates: First submitted 2020-01-27; First posted 2020-04-24 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2020-01

CONDITIONS: Vaginal Disease
MeSH Terms: conditions — Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: Post Marketing Follow Up Study.
  Enrolled patients will be 75, divided as follows:
  * 25 patients belonging to study DMS/18/AINARA/01 (only Arm A, Ainara®)
  * 50 patients belonging to study DMS/18/AINARA/02
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ainara (Experimental): Ainara is a class II medical device, already marketed in several EU countries. The product is a mucoadhesive moisturising gel for vulvovaginal use, indicated for the relief of symptoms of vaginal atrophy and dryness, and related discomfort. In each packaging there is a tube containing the gel (sterile and viscous with about 87% water) and a syringe-like plastic applicator with cannula and plunger.
  Each administration kit (subject kit) for patients of Ainara® will contain a box with 1 tube with 30 g gel, 1 cannula and 1 plunger. The gel quantity is enough for one subject over the course of the study (1 g at each administration).
  Interventions: Device: Ainara

INTERVENTIONS:
Device: Ainara — 1 g at each administration

SUMMARY:
The objective of the present PMCF study with a 6 month follow up period is to identify potential new and unknown risks associated with longer term use of Ainara® and (considering the duration of symptoms in GSM) to collect additional data regarding efficacy of a long-term treatment with this medical device.

DETAILED DESCRIPTION:
This is an interventional prospective study. It fits/pertains into the category of Post Marketing Clinical Follow up studies. The study evaluates performance, safety, and quality of life in late menopausal transition and post-menopausal women treated with the medical device Ainara® vaginal gel for vaginal dryness for 6 months The Research Question of the present study is the following: in a population composed of menopausal transition and menopausal women treated with polycarbophilic vaginal gel (Ainara®) for vaginal dryness, will a 6-month post marketing follow up study be able to give a reliable overview on the long-term performance (in terms of VHI, subjective and objective symptoms, and female sexual function), safety (in terms of patient and Investigator evaluation, and potential unknown risks of ADE/SADE/USADE/AE/SAE) and quality of life of this medical device.

ELIGIBILITY:
Inclusion Criteria:

1. Women previously treated with Ainara® vaginal gel in the study DMS/18/AINARA/01 or DMS/18/AINARA/02.
2. Non-pregnant and in late menopausal transition (with a break in menstrual periods of at least 60 days), or post-menopausal (total cessation of menses for ≥ 1 year) women following STRAW criteria and considering the screening date of the study (DMS/18/AINARA/01 or DMS/18/AINARA/02) in which they were enrolled.
3. Women aged ≥ 45 to ≤ 70 years (considering the baseline date of the study DMS/18/AINARA/01 or DMS/18/AINARA/02 in which they were previously enrolled);
4. Body mass index (BMI) ≥ 18.5 to ≤ 36 kg/m2
5. Females of childbearing potential who agree to use only lubricated condoms or spiral as contraceptives methods, during the full duration of the study.
6. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.
7. Capable of and freely willing to provide written informed consent prior to participating in the study.

Exclusion Criteria:

Subjects fulfilling one or more of the following exclusion criteria will NOT be included in the study:

1. Malignancy (also leukemic infiltrates) within 5 years prior to Day 1 (except for treated basal cell/squamous cell carcinoma of the skin).
2. Genital bleeding.
3. Estrogen vaginal treatment during the study period (it was permitted only if terminated at least 6 months before study).
4. Systemic estrogen therapy (it was permitted only if terminated at least 6 months before study).
5. Subjects with illness, or other medical condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the study.
6. Clinical evidence of acute infection currently requiring treatment (syphilis, herpes simplex, human papilloma virus, gonorrhea, chlamydia, lymphogranuloma venereum, etc.); clinical evidence or history of chronic infectious disease (i.e. tuberculosis).
7. Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt or suicidal ideation, or any other psychiatric illness (except for intermittent anxiety).
8. Known allergy to tested IMDs or its excipients.
9. Drug or alcohol abuse 12 months prior to Day 1.
10. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days (except DMS/18/AINARA/01 or DMS/18/AINARA/02).
11. Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female subjects can have a vaginal disease
Enrollment: 73 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Vaginal Health Index (VHI) | 180 days
  To measure the Ainara®'s efficacy on vaginal dryness the same outcomes used in the two trials DMS/18/AINARA/01 and DMS/18/AINARA/02 were chosen: Vaginal Health Index (VHI) by Investigator. For outcome the change from baseline to Visit 2 (final visit) will be analyzed; Minimal value for VHI is 1 and maximal value for VHI is 5. A higher score on VHI means an improvement in vaginal health
Visual Analogue Scale (VAS) for vaginal dryness evaluated by subjects | 180 days
  To measure the Ainara®'s efficacy on vaginal dryness the same outcomes used in the two trials DMS/18/AINARA/01 and DMS/18/AINARA/02 were chosen: the Visual Analogue Scale (VAS) by the subject. For the VAS outcome the change from baseline to Visit 2 (final visit) will be analyzed; in addition, VAS mean value will be compared with the value at days 30, 60, 90, 120, and 150.
SF 12 questionnaire completed by the patient | 180 days
  Quality of Life will be evaluated by SF12 questionnaire, a binary (Yes/No) and multiple choice-type survey, widely used to assess general health. Data will be analyzed comparing scores from baseline visit to Visit 2 (final visit).
ADE/SADE/USADE (adverse device event, serious adverse device event unexpected serious device event) and AE/SAE | 180 days
  Safety will be evaluated by the collection of ADE/SADE/USADE (adverse device event, serious adverse device event unexpected serious device event) and AE/SAE, • ADE/SADE/USADE and AE/SAE; Patient Global evaluation of safety (PGAS); Investigator Global evaluation of safety (IGAS);

SECONDARY OUTCOMES:
Rate of subjective symptoms | 30, 60, 90, 120, 150, 180 days
  subjective symptoms: dryness, itching, burning, dyspareunia, and dysuria reported on patient diary and scored as reported in the AGATA study as follows: 0 = absence, 1 = slight, 2 = moderate, and 3 = severe intensity. The change in these variables will be evaluated from baseline to days 30, 60, 90, 120, 150, and 180 (final visit).
Objective signs in vaginal mucosa | 180 days
  Objective signs in vaginal mucosa: dryness, thinning rugae, pallor, fragility, and petechiae evaluated by Investigator as: 0 = absence, 1 = slight, 2 = moderate, and 3 = severe alteration. The change in these variables will be evaluated from baseline to Visit 2 (final visit).
Vaginal pH | 180 days
  Vaginal pH: it will be measured by the Investigators with a test strip delivered by Sponsor. The baseline values can be from 5.0 (this was the minimum value need for vaginal atrophy diagnosis in AGATA study) to 9.0. The Investigator will insert the pH strip into the upper wall of the vagina and will consider the reading made while the strip is still damp. For this outcome the change of mean values will be analysed from baseline to Visit 2 (final visit).
Global Symptom Score (GSS) | 180 days
  Global Symptom Score (GSS)(20) a composite score of symptoms, will be obtained to assess the effect of treatment on all individual symptoms taken as a whole. It will be calculated by the addition of the intensity scores of all individual symptoms (range, 1-15: 1 = only mild vaginal dryness, 15 = all five symptoms severe in intensity). This outcome will be analysed assessing the change from baseline visit to day 180 visit (final visit).
Female Sexual Function Index (FSFI) | 90, 180 days
  Female Sexual Function Index (FSFI) Romanian version, evaluated by Investigator and analysed considering the change from baseline to 90 and 180 days (final visit). The minimum score of this scale is 19 and the maximum value is 95. A higher score means an improvement in sexual function of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Liviu Cristian Patrascu, MD, Principal Investigator — Fizio Center
Locations (1):
- Fizio Center, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No